CLINICAL TRIAL: NCT06811194
Title: Prospective Cohort Study of Prior Myocardial Infarction Identification on Electrocardiogram: the PRIME Cohort Study
Brief Title: PRIor Myocardial Infarction Identification on Electrocardiogram
Acronym: PRIME
Status: Enrolling by invitation | Type: Observational
Sponsor: The Third People's Hospital of Chengdu (Other)
Responsible Party: Principal Investigator, Hanxiong Liu, Principal Investigator, The Third People's Hospital of Chengdu
Other Study IDs: Third Hospital Chengdu
Record Dates: First submitted 2025-01-22; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Prior Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Paper records include symptoms, signs, events, and electrocardiograms (ECGs)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Multicenter Cohort Study of Prior Myocardial Infarction: Myocardial infarction is a disease that affects the heart muscle, leading to a reduction in its function. When a patient has experienced a myocardial infarction in the past but no longer exhibits acute symptoms, it is referred to as an old myocardial infarction. This condition is typically characterized by the scarring of heart muscle tissue, resulting in partial loss of cardiac function. Patients may develop complications such as heart failure and arrhythmias. Although the symptoms may be mild, regular monitoring of cardiac function and status is essential. Early detection and management can effectively prevent further cardiovascular events. Therefore, regular medical check-ups and adherence to medical advice are crucial. For patients with a history of myocardial infarction, lifestyle modifications and pharmacological therapy are also important components in the recovery and maintenance of cardiac health.

SUMMARY:
Abstract Background: Chronic myocardial infarction (MI) is a serious cardiovascular disease associated with high mortality rates, making early diagnosis and timely intervention essential for improving patient outcomes. However, some patients may present without clear symptoms or relevant medical histories, complicating the diagnostic process. Currently, diagnosis predominantly relies on electrocardiograms (ECGs) and imaging tests. Although cardiac magnetic resonance imaging (MRI) is regarded as the gold standard, its high cost and complexity hinder its clinical application. Consequently, there is an urgent need for new ECG diagnostic criteria to mitigate the risks of misdiagnosis and missed diagnoses.

Objective: This study aims to explore new diagnostic criteria to enhance the accuracy of ECG diagnoses for chronic MI.

Methods: This research is a prospective, multicenter cohort study designed to assess the impact of newly developed ECG diagnostic criteria on the accuracy of chronic myocardial infarction (MI) diagnoses. The study spans a 60-month period, including a 12-month patient enrollment phase. Participants will comprise individuals aged 35 to 85 who meet the inclusion criteria: those diagnosed with chronic myocardial infarction via ECG, those with a definitive history of MI (≥3 months), or individuals clinically suspected of having coronary artery disease with at least two coronary risk factors. Data collection will include clinical symptoms, signs, ECG findings, and cardiac magnetic resonance (CMR) findings, the latter serving as a primary endpoint. Follow-up will focus on changes in patients' symptoms and ECG assessments. Statistical analysis software will be employed to evaluate the influence of the new diagnostic criteria on rates of missed and misdiagnosis.

DETAILED DESCRIPTION:
Abstract Background: Chronic myocardial infarction (MI) is a serious cardiovascular disease associated with high mortality rates, making early diagnosis and timely intervention essential for improving patient outcomes. However, some patients may present without clear symptoms or relevant medical histories, complicating the diagnostic process. Currently, diagnosis predominantly relies on electrocardiograms (ECGs) and imaging tests. Although cardiac magnetic resonance imaging (MRI) is regarded as the gold standard, its high cost and complexity hinder its clinical application. Consequently, there is an urgent need for new ECG diagnostic criteria to mitigate the risks of misdiagnosis and missed diagnoses.

Objective: This study aims to explore new diagnostic criteria to enhance the accuracy of ECG diagnoses for chronic MI.

Methods: This research is a prospective, multicenter cohort study designed to assess the impact of newly developed ECG diagnostic criteria on the accuracy of chronic myocardial infarction (MI) diagnoses. The study spans a 60-month period, including a 12-month patient enrollment phase. Participants will comprise individuals aged 35 to 85 who meet the inclusion criteria: those diagnosed with chronic myocardial infarction via ECG, those with a definitive history of MI (≥3 months), or individuals clinically suspected of having coronary artery disease with at least two coronary risk factors. Data collection will include clinical symptoms, signs, ECG findings, and cardiac magnetic resonance (CMR) findings, the latter serving as a primary endpoint. Follow-up will focus on changes in patients' symptoms and ECG assessments. Statistical analysis software will be employed to evaluate the influence of the new diagnostic criteria on rates of missed and misdiagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 35 and 85 years.
* Patients must meet at least one of the following conditions:

  * Diagnosis of prior MI based on ECG (as per the fourth universal definition of MI).
  * History of prior MI (≥3 months post-MI).
  * Any clinical suspicion of coronary artery disease (CAD) with at least two of the following risk factors:

Male age >50 years or female age >60 years. Diabetes mellitus. Hypertension. Hypercholesterolemia requiring medication. Family history of premature CAD (first-degree relatives: male ≤55 years, female ≤65 years).

Body mass index (BMI) ≥30 kg/m². History of peripheral vascular disease. History of coronary artery intervention or bypass surgery. Informed consent obtained

Exclusion Criteria:

* Life expectancy <1 year due to non-cardiovascular diseases.
* Contraindications to cardiac MRI or inability to complete the examination.
* History of non-ischemic cardiomyopathy.
* History of heart transplantation.
* Acute MI within the past 30 days.
* During pregnancy.

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: An old MI is a condition in which the patient has experienced a myocardial infarction in the past, but no acute symptoms are present at this time. This condition usually manifests as scarring of the heart muscle tissue, resulting in a partial loss of heart muscle function. Patients may experience complications such as heart failure and arrhythmia, and although the symptoms may be mild, it is still necessary to regularly monitor the function and status of the heart. Early detection and management can effectively prevent further cardiovascular events, so regular medical check-ups and following medical advice are particularly important. For patients who have had an old heart attack, lifestyle adjustments and medication are also important components of restoring and maintaining heart health
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2025-02-20 (Estimated); Primary Completion 2026-02-20 (Estimated); Study Completion 2031-02-20 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular death or nonfatal MI. | 60 Months after Enrollment
  Primary outcome: cardiovascular death or nonfatal MI occurred during the 60-month follow-up after enrollment.

SECONDARY OUTCOMES:
A composite of cardiovascular death, nonfatal MI, hospitalization for unstable angina or congestive heart failure, and late unplanned CABG. | 60 Months after Enrollment
  Secondary outcome was defined by a composite of cardiovascular death, nonfatal MI, hospitalization for unstable angina or congestive heart failure, and late unplanned CABG.

CONTACTS AND LOCATIONS:
Locations (1):
- The Third People's Hospital of Chengdu, Chengdu, Sichuan, China